CLINICAL TRIAL: NCT02934789
Title: Randomized Prospective Study of the Effectiveness of the Truclear Device for Hysteroscopic Myomectomy on Patient Quality of Life
Brief Title: Effectiveness of Truclear on Patient Quality of Life
Acronym: HSCMyomecty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All For Women Healthcare, Illinois (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2015-17
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Heavy Menstrual Bleeding
Keywords: submucosal fibroids; heavy menstrual bleeding; quality of life
MeSH Terms: conditions — Menorrhagia | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group: surgical arm (Active Comparator): Hysteroscopic myomectomy with Truclear done on patients with abnormal uterine bleeding and submucosal fibroid(s).
  Interventions: Procedure: Hysteroscopic myomectomy with Truclear
- Control group: medical arm (Active Comparator): Medical therapy for patients with abnormal uterine bleeding/ heavy menses and submucosal fibroids
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Procedure: Hysteroscopic myomectomy with Truclear — Hysteroscopic myomectomy with Truclear done on patients with abnormal uterine bleeding and submucosal fibroid(s).
  Other Names: Truclear
  Arms: Study group: surgical arm
Drug: Medical therapy — Medical therapy for patients with abnormal uterine bleeding/ heavy menses and submucosal fibroids.
  Other Names: oral contraceptive pills, Mirena intrauterine device
  Arms: Control group: medical arm

SUMMARY:
This study aims to evaluate the quality of life in patients treated for submucosal leiomyomas using the Truclear hysteroscopic morcellator compared to women managed medically. Study population includes women age 18 and older with symptomatic submucosal myomas. Patients will be asked to complete the Uterine Myoma Symptom and Health-related Quality of Life Questionnaire (UFS-QOL) at enrollment and at 1, 3, and 6 months after treatment.

DETAILED DESCRIPTION:
Submucosal myomas are a common cause of pelvic complaints and abnormal uterine bleeding (AUB) and there are many available modalities for treatment. Hysteroscopic myomectomy is a minimally invasive approach for removal of submucosal leiomyomas. Alternatively, medical management can be attempted. This study aims to evaluate the quality of life in patients treated for submucosal leiomyomas using the Truclear hysteroscopic morcellator compared to women managed medically. Study population includes women age 18 and older with symptomatic submucosal myomas. Patients will be asked to complete the Uterine Myoma Symptom and Health-related Quality of Life Questionnaire (UFS-QOL) at enrollment and at 1, 3, and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abnormal uterine bleeding and submucosal fibroid(s) undergoing hysteroscopic myomectomy or medical therapy with oral contraceptive pills
* Patients with Type 0, 1 or 2 submucosal myomas

Exclusion Criteria:

* Pregnant women
* Patients with suspicion of uterine malignancy
* Patients without submucosal fibroid seen during planned hysteroscopic myomectomy
* Patients with active vaginal infection
* Patients with contraindication to hysteroscopic myomectomy
* Patients with cognitive impairment who are unable to provide consent and adequately complete the questionnaire.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-09; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Quality of life score | Two years
  Primary outcome is the health-related quality of life (HR-QOL) as reflected from UFS-QOL scores.

SECONDARY OUTCOMES:
Secondary surgical outcomes | Two years
  Secondary surgical outcomes include estimated blood loss (EBL), operating time (OT), pedal resection time, fluid deficit, total fluid use, pathology report (including total myoma weight), surgical outcome and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Tam, MD, Principal Investigator — All For Women Healthcare
Locations (1):
- All For Women Healthcare, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Spies JB, Bradley LD, Guido R, Maxwell GL, Levine BA, Coyne K. Outcomes from leiomyoma therapies: comparison with normal controls. Obstet Gynecol. 2010 Sep;116(3):641-652. doi: 10.1097/AOG.0b013e3181ed36b3. PMID 20733447